CLINICAL TRIAL: NCT06456112
Title: Construction and Validation of a Diagnostic Model for Predicting Molecular Residual Disease and Recurrence of Cervical Cancer Based on Circulating Tumor HPV
Status: Not yet recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: YingZhou 2024-7
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Systematic evaluation of the value of molecular residual lesions of cervical cancer based on circulating tumor HPV in the prognostic evaluation and recurrence monitoring of cervical cancer patients.

DETAILED DESCRIPTION:
Cervical cancer has a very clear etiology, with the vast majority of cases being caused by persistent and repeated infections with high-risk HPV. In the carcinogenic mechanism of cervical cancer, there are large amounts of HR-HPV integrated into the human genome in cancer cells; these HR-HPV can be released into the bloodstream in the form of ctHPV, and most patients with stages I-IV of cervical cancer can have detectable ctHPV in their blood. Among them, the detection rate in the blood of late-stage patients ranges from 63.3% to 100%. Several studies have demonstrated that ctHPV may serve as a marker for monitoring recurrent tumor molecular residual lesions, which could be of significant importance for prognostic evaluation and monitoring whether the disease has recurred. In this study, we will systematically evaluate the value of molecular residual lesions of cervical cancer based on circulating tumor HPV in the prognostic evaluation and recurrence monitoring of cervical cancer patients

ELIGIBILITY:
Inclusion Criteria:

1. Women, aged between 18 and 75 years, can receive standard treatment, including patients who only receive surgery, and patients who receive radiotherapy and chemotherapy after surgery.
2. Cervical cancer caused by HPV16 or HPV18 infection diagnosed by molecular biology or pathological tissue (p16), with pathological stage of IB1 to IV.

   -

Exclusion Criteria:

1. Patients with other malignancies
2. Patients with any uncontrolled systemic disease, including active infection, uncontrolled hypertension, diabetes mellitus, unstable angina and congestive heart failure, myocardial infarction (1 year) before starting treatment, severe arrhythmia requiring medical treatment, coagulation abnormalities, liver or kidney or metabolic disease
3. Cervical cancer patients who had undergone LEEP knife or conization in primary hospitals
4. Cervical cancer patients whose peripheral blood was negative for ctHPV at baseline. Here, ctHPV negative refers to patients who are both negative for ddPCR and NGS

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cervical cancer patients diagnosed with HPV16 or HPV18 infection
Sampling Method: Non-Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
The one-year probability of OS | one year
  OS (overall survival) is defined as the time which begins at diagnosis and up to the time of death

SECONDARY OUTCOMES:
PFS | 1 month post treatment
  progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zhou, MD, Study Chair — The First Affiliated Hospital of USTC (Anhui Provincial Hospital)
Locations (1):
- Anhui Provincal Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No